CLINICAL TRIAL: NCT04162301
Title: A Phase I, Open-Label, Multiple-Dose, Dose Escalation and Expansion Study to Investigate the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activities of CS3002, a CDK4/6 Inhibitor, in Subjects With Advanced Solid Tumors
Brief Title: A Study of CS3002 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study has been stopped for strategic and business reasons.
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CS3002-101
Record Dates: First submitted 2019-10-29; First posted 2019-11-14 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS3002 CDK4/6 inhibitor (Experimental)
  Interventions: Drug: CS3002

INTERVENTIONS:
Drug: CS3002 — CS3002 tablet will be orally administered daily for 3 weeks followed by 1 week off treatment, defining a treatment cycle of 28 days in duration.

SUMMARY:
This is a phase I, open-label, multiple-dose, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics and anti-tumor activity of CS3002 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject or a legally acceptable representative has been informed of all pertinent aspects of the study.
2. Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
3. Male or female and ≥ 18 years of age on the day of signing informed consent.
4. Subjects with histologically or cytologically confirmed metastatic or locally advanced unresectable solid tumor (except SCLC and HPV positive tumors), who has experienced disease progression following treatment with all available standard therapy, or for whom treatment is not available, not tolerated or refused.
5. Subjects with at least one measurable lesion as defined per RECIST v1.1 (only bone metastasis or CNS as measurable focus is not allowed).
6. ECOG performance status ≤ 1.
7. Able to swallow and retain oral medication.
8. Subject must have adequate organ function as indicated by the following laboratory values, under the circumstance of not receiving blood transfusion, EPO, Granulocyte Colony-Stimulating Factor (G-CSF) or other medical support within 14 days before study drug administration
9. Non-pregnant and non-nursing. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to the first dose of CS3002 (WOCBP is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 months). WOCBP must agree to remain abstinent (refrain from heterosexual intercourse) or use an acceptable contraceptive method (refer to Appendix 6) from the day of signing informed consent, during the treatment period and for at least 90 days after the last dose of study drug.
10. Men must agree to remain abstinent (refrain from heterosexual intercourse) or use an acceptable contraceptive method (refer to Appendix 6) from the day of signing informed consent, during the treatment period and for at least 90 days after the last dose of study drug. Men must refrain from donating sperm during this same period.
11. (Part 2 only) Subjects must provide the most recent available sample containing adequate formalin-fixed paraffin-embedded (FFPE) tumor-derived material (tumor blocks or 3 slides minimum) from a core needle biopsy or surgery for analysis of biomarkers, and willing to accept on-treatment biopsy as scheduled in protocol.

Exclusion Criteria:

1. Prior treatment with any CDK4/6 inhibitor.
2. Participation in other studies involving investigational drug(s) within 28 days prior to the first dose of CS3002 and/or during study participation.
3. Acceptance of major surgery, chemotherapy, radiotherapy, target therapy, immunotherapy or other anti-cancer therapy within 21 days prior to the first dose of CS3002.
4. Prior treatment with drugs that are known to prolong the QT interval within 7 days before the first dose of CS3002.
5. Concomitant use of products known to prolong the QT interval or to be moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued ≥ 5 half-lives prior to first dose of CS3002 and withheld throughout the trial until 2 weeks after the last dose of CS3002.
6. Any toxic effects of prior anti-cancer therapy or surgical procedures unresolved to baseline severity or NCI-CTCAE Version 5.0 Grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion)
7. Diagnosis of any other malignancy within 3 years prior to the first dose of CS3002, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
8. Diagnosis of small cell lung cancer and HPV positive tumors.
9. Known brain metastasis or other central nervous system (CNS) metastasis that is either symptomatic or untreated. CNS metastases that have been treated by complete resection and/or radiotherapy demonstrating stability or improvement are not an exclusion criterion provided they are stable as shown by imaging for at least 4 weeks before screening without evidence of cerebral edema and no requirements for corticosteroids or anticonvulsants.
10. History of allergic reactions attributed to compounds of similar chemical or biologic composition to CS3002, or any of its excipients (refer to Section 6.2.1).
11. Patients with advanced, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term (including patients with massive uncontrolled effusions [pleural, pericardial, peritoneal], and pulmonary lymphangitis).
12. Any of the following within 6 months prior to the first dose of CS3002: myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of NCI-CTCAE Version 5.0 Grade ≥ 2, atrial fibrillation of any grade, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident including transient ischemic attack, or symptomatic pulmonary embolism.
13. Presence of active gastrointestinal disease or other condition that will impair significantly with the absorption, distribution, metabolism, or excretion of CS3002.
14. Uncontrolled intercurrent illness including, but not limited to, known ongoing or active infection, including HIV, active hepatitis B or C.
15. Subjects who are Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) positive, or Hepatitis C virus (HCV) antibody positive at screening, must not be enrolled until further definite testing with Hepatitis B virus (HBV) DNA titres and HCV RNA tests can conclusively rule out presence of active infection (HBV DNA ≥1000 cps/mL or 200 IU/mL; HCV RNA exceeding the lower detection limit) requiring antiviral therapy with Hepatitis B and C, respectively.
16. QTc interval > 480 msec (based on the mean value of the triplicate screening ECG); family or personal history of long or short QT syndrome; history of ventricular dysrhythmias or risk factors for ventricular dysrhythmias such as structural heart disease (e.g., severe left ventricular systolic dysfunction, left ventricular hypertrophy), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia).
17. Known or suspected active alcohol or drug abuse.
18. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
19. Females who are pregnant or lactating.

For more information regarding trial participation, please contact at cstonera@cstonepharma.com

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v5.0 | Subjects will be monitored for safety and tolerability throughout the study until 30 ±3 days since the last dose of investigational product or until initiation of a new anti-cancer treatment, whichever occurs first.
  incidence rate and characteristics of dose-limiting toxicity (DLT); incidence and severity of adverse events (AEs) and serious adverse events (SAEs), including changes of laboratory values, vital signs and electrocardiogram (ECG) findings. And based on the safety, tolerability, pharmacokinetics, preliminary efficacy, and other available data to determine MTD, RP2D and regimen for CS3002.

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Huang, Study Director — CStone Pharma
Locations (2):
- Australia (2):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Peninsula and South Eastern Haematology and Oncology Group, Heidelberg, Victoria